CLINICAL TRIAL: NCT05559502
Title: Comparison of High Flow Nasal Oxygenation Versus Endotracheal Intubation on Recovery Profiles in Laryngeal Microsurgery
Brief Title: High Flow Nasal Oxygenation vs Endotracheal Intubation on Recovery Profiles in Laryngeal Microsurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJOUIRB-IV-2022-457
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cough
Keywords: High flow nasal oxygenation; Laryngeal microsurgery; emergence cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNO group (Experimental): Patients will receive HFNO therapy during laryngomicrosurgery.
  Interventions: Device: HFNO group
- ET group (Active Comparator): Endotracheal intubation was performed for general anesthesia
  Interventions: Device: ET group

INTERVENTIONS:
Device: HFNO group — HFNO therapy make possible to perform tubeless anesthesia, providing perfect exposure of structure of the vocal cords.
  Other Names: Optiflow
  Arms: HFNO group
Device: ET group — Endotracheal tube is a plain tube, which is most commonly used in general anesthesia.
  Other Names: Portex, Smiths Medical International Ltd., South East England, United Kingdom
  Arms: ET group

SUMMARY:
Transnasal humidified rapid-insufflation ventilatory exchange(THRIVE), or also termed high flow nasal oxygenation (HFNO) is a method of supplying heated, humidified high concentrations of oxygen via nasal cavity. This study hypothesizes that in general anesthesia for laryngeal microsurgery, high-flow nasal oxygen without endotracheal intubation reduces cough during the emergence period compared to endotracheal intubation.

DETAILED DESCRIPTION:
Laryngeal microsurgery is mainly performed by a conventional method of general anesthesia with endotracheal intubation (ET), which may have difficulty accessing the lesion behind the larynx, and may be limited in securing space for surgical manipulation. To compensate for these shortcomings, a method of maintaining general anesthesia without using an endotracheal tube has been introduced, and high-flow nasal oxygen(HFNO) and transnasal humidified rapid insufflation ventilatory exchange(THRIVE) enable tubeless anesthesia due to apnea oxygenation and apnea ventilation effect during laryngeal microsurgery. Coughing and straining can be accompanied by emergence after general anesthesia. Forceful vocal cord adduction especially after upper respiratory surgery such as laryngeal microsurgery can cause damage and bleeding of surgical tissue, delaying wound healing. If a small amount of remifentanil is continuously injected during emergence after total intravenous anesthesia(TIVA), airway complications such as coughing can be reduced during emergence without delay in recovery time, and hemodynamic stability can be promoted. In this study, the effect of endotracheal intubation and high-flow nasal oxygen on the emergence cough and postoperative sore throat is compared when total intravenous anesthesia(TIVA) using propofol and remifentanil is performed in patients undergoing laryngeal microsurgery. This study hypothesizes that in general anesthesia for laryngeal microsurgery, high-flow nasal oxygen without endotracheal intubation reduces cough during the emergence period compared to endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists classification 1 or 2 who receive general anesthesia for laryngeal microsurgery

Exclusion Criteria:

* Patients with major cardiovascular, pulmonary, and cerebrovascular disease
* Laser laryngeal surgery
* Morbid obesity (BMI>35 kg/m2)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Grade of Emergence cough during periextubation period | From end of surgery to extubation
  Grade Score (grade 0=no cough, grade 1=light or single cough, grade 2=moderate cough or more than one episode of nonsustained coughing, grade 3=sustained and repetitive cough movements with head lift, 0 is the minimum value which is a better outcome and 3 is the maximum value which is a worse outcome.)

SECONDARY OUTCOMES:
Number of Participants with postoperative airway complications | from 1 hour after surgery to 24 hours after surgery
  post operative sore throat

CONTACTS AND LOCATIONS:
Overall Officials: JongYeop Kim, M.D.,Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeongki-do, South Korea